CLINICAL TRIAL: NCT04868201
Title: A Self-guided App-Based Virtual Reality Cognitive Behavior Therapy for Anxiety Disorder in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Laiana A. Quagliato, MD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 74646917.1.0000.5263
Record Dates: First submitted 2021-04-25; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Anxiety Disorders
Keywords: anxiety; virtual reality; app; self-guided; Cognitive behavior therapy
MeSH Terms: conditions — Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0-anxiety (Experimental): 0-anxiety is based on the principles of VRT and CBT, which currently is the most researched and used treatment for anxiety disorders. The 0-anxiety intervention is an app-based intervention consisting of six modules that can be followed according to a user's own timing and without the intervention of a therapist.
  Interventions: Device: 0-anxiety
- wait-list condition (No Intervention)

INTERVENTIONS:
Device: 0-anxiety — 0-anxiety is a self-guided app-based utilizing virtual reality establish in cognitive behavior therapy treatment.
  Arms: 0-anxiety

SUMMARY:
To examine the efficacy of a fully self-guided app-based virtual reality cognitive behavior therapy (VR CBT) using low-cost (cardboard) virtual reality goggles compared with a wait-list control group and to determine its user friendliness. We hypothesize that children with GAD enrolled in the self-guided app will present lower scores of anxiety.

DETAILED DESCRIPTION:
A randomized controlled design will be carried out, in which the effectiveness and user- friendliness of an online app-based VR self-help treatment '0-anxiety' will be evaluated. Our primary objective is to determine the clinical effects (a reduction in anxiety symptoms at post-test [between the experimental condition and controls] of 0-anxiety, and whether effects are sustainable at follow-up [a reduction in anxiety symptoms between baseline and follow-up for those in the experimental condition]). Our secondary objective is to determine the user-friendliness of 0-anxiety. In this study, 230 children from the Brazilian population will be randomized over 2 conditions: the experimental condition (0-anxiety) and a waitlist condition. The duration of the intervention will be 3 weeks. Measures will be taken at baseline, directly after the intervention (3 weeks) and at 3 months (follow-up). All measures will be completed online. Therefore, the child will participate in the study in his/her natural environment. Subjects in the wait-list condition will receive the intervention after completion of the post-test. Randomization (block-randomization) will be performed by an independent researcher.

ELIGIBILITY:
Inclusion Criteria:

* individuals must be between 8-12 years old;
* subjects must score above 25 on the SCARED questionnaire;
* subjects must have access to a smart phone and internet;
* individuals must be willing to participate in the research study and providing informed consent.

Exclusion Criteria:

* children that present with symptoms of severe depression or suicidality as measured with KSADS-PL26;
* children that have insufficient knowledge of the Portuguese language;
* subjects that are under any current treatment for anxiety disorder or using psychotropic medication.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels | baseline and and 3 months after the completion of the intervention
  Screen for Child Anxiety Related Disorders (SCARED). A score above 25 indicates a significant level of anxiety. Higher scores mean worse anxiety levels.

SECONDARY OUTCOMES:
Fear Survey Schedule for Children-Revised (FSSC-R) | baseline, 3 weeks after the intervention, and 3 months after the completion of the intervention
  The FSSC-R is a widely used self-report measure of children and adolescents' fears. The instrument, a revision of Scherer and Nakamura's (1968) original Fear Survey Schedule for Children, contains 80 items that are each rated on a three-point scale (none, some, a lot). A total fearfulness score can be obtained, as can five subscale scores based on a factor analysis of the items. In addition, the number of intense fears can be indicated (i.e., the number of fears endorsed 'a lot'), as can the most prevalent fears for a given child/adolescent or group of children and adolescents (i.e., boys, preadolescents, school phobic youngsters, etc.). Higher scores mean worse fear levels.
Spence Children's Anxiety Scale - Parent and Children version | baseline, 3 weeks after the intervention, and 3 months after the completion of the intervention
  The scale is completed by a parent of an anxious child between the ages of 6 to 18. It provides an overall measure of anxiety together with scores on six sub-scales each tapping a specific aspect of child anxiety. - Panic attack and agoraphobia - Separation anxiety - Physical injury fears - Social phobia - Obsessive compulsive - Generalized anxiety disorder / overanxious disorder. This yields a maximum possible score of 114. Higher scores mean worse anxiety levels.

IPD SHARING:
Plan to Share IPD: Undecided